CLINICAL TRIAL: NCT06064656
Title: Clinical Characteristics and Mortality in Patients With Fibrodysplasia Ossificans Progressiva (FOP): A Non-Interventional US National Retrospective Cohort
Brief Title: A Non-Interventional Study of Clinical Characteristics and Mortality of US Patients With Fibrodysplasia Ossificans Progressiva (FOP)
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R2477-FOP-2143
Record Dates: First submitted 2023-09-11; First posted 2023-10-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Fibrodysplasia Ossificans Progressiva (FOP)
Keywords: Genetic disease; Heterotopic ossification (HO); Skeletal dysplasia; Activin A receptor, type I (ACVR1)
MeSH Terms: conditions — Myositis Ossificans; Genetic Diseases, Inborn; Ossification, Heterotopic; Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FOP Cohort: Sub-Cohort 1: All patients with active enrollment (closed claims) during part or all the study period (2018-2023) Sub-Cohort 2: All patients with both active enrollment (closed claims) and open claims encounters during study period (2018-2022)
  Interventions: Other: Non-Interventional
- Comparator Cohort: All individuals without FOP and with active enrollment (closed claims) during part or all of the study period (2018-2023)
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — No study treatment will be administered in this study.

SUMMARY:
Primary Objective(s):

* To describe the demographic characteristics of people living with FOP and a matched cohort of non-FOP people living in the United States (U.S.)
* To describe the prevalence of clinical characteristics of interest and the use of key medications in people living with FOP and a matched cohort of non-FOP people living in the U.S.
* To compare the prevalence of key clinical characteristics and medication use in people living with FOP to a matched cohort of non-FOP people living in the U.S.
* To estimate the crude mortality rate among people living with FOP

ELIGIBILITY:
Inclusion Criteria:

FOP Cohort(s):

1. Living with FOP in the United States who have been identified from the IFOPA membership database
2. Confirmed FOP diagnosis through IFOPA membership database will be tokenized and linked with HealthVerity's medical claims data, pharmacy claims data, laboratory data and obituary data, as defined in the protocol

Comparator Cohort:

1. People without FOP living in the U.S. randomly sampled from HealthVerity's closed medical claims data and matched to the FOP population
2. Index date are defined as each person's cohort entry date. People may exit and re-enter the cohort, with the period during which they were not in the cohort excluded from the analysis
3. The comparator cohort will be matched to the cohort of people with FOP on the following variables: age, sex, insurance type and first index date

Exclusion Criteria:

1. Failure to meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: FOP Cohort(s):
  The International Fibrodysplasia Ossificans Progressiva Association (IFOPA) membership has 235 confirmed people living with FOP in the US. From this membership database, there were 131 members or next of kin of members who opted-in to allow for the tokenization of their membership data to occur.
  Comparator Cohort:
  A random sample of 100,000 people from an insured population without FOP diagnosis living in the U.S. and matched to the FOP population.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics | Up to 5 years
Prevalence of cardiovascular disease | Up to 5 years
Prevalence of metabolic disease | Up to 5 years
Prevalence of hematology disease | Up to 5 years
Prevalence of infection | Up to 5 years
Prevalence of respiratory disease | Up to 5 years
Prevalence of reproductive disease | Up to 5 years
Prevalence of neurologic disorders | Up to 5 years
Prevalence of skeletal disorders | Up to 5 years
Prevalence of gastrointestinal disease | Up to 5 years
Prevalence of hearing loss | Up to 5 years
Prevalence of dermatologic disorders | Up to 5 years
Prevalence of neoplasms | Up to 5 years
Average number of dispensations per FOP patient per year | Up to 5 years
Cumulative number of dispensations per FOP patient | Up to 5 years
Incidence of all-cause death | Up to 5 years
  FOP Sub-Cohorts 1 and 2 Only

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron, Tarrytown, New York, United States